CLINICAL TRIAL: NCT04866446
Title: Evaluation of The Effects of Personal Protective Equipment During Airway Management; A Prospective, Non-randomized, Controlled, Simulation Study
Brief Title: Evaluation of The Effects of Personal Protective Equipment During Airway Management
Status: Completed | Type: Observational
Sponsor: Kezban Aydan Okuyucu (Other)
Responsible Party: Sponsor-Investigator, Kezban Aydan Okuyucu, Medical Doctor, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Other Study IDs: derinceanesteziaydan-1
Record Dates: First submitted 2021-01-06; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Personal Protective Equipment; Airway Management
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal airway manikin with standard uniform: The participants will carry out intubation procedure using macintosh direct laryngoscope, GlideScope video laryngoscope, C-Mac video laryngoscope and Frova intubation catheter and laryngeal mask insertion using ProSeal LMA and I-gel LMA, respectively.
  Interventions: Device: endotracheal intubation and laringeal mask airway insertion
- normal airway manikin with personal protective equipment: The participants will carry out intubation procedure using macintosh direct laryngoscope, GlideScope video laryngoscope, C-Mac video laryngoscope and Frova intubation catheter and laryngeal mask insertion using ProSeal LMA and I-gel LMA, respectively.
  Interventions: Device: endotracheal intubation and laringeal mask airway insertion
- difficult airway manikin with standard uniform: The participants will carry out intubation procedure using macintosh direct laryngoscope, GlideScope video laryngoscope, C-Mac video laryngoscope and Frova intubation catheter and laryngeal mask insertion using ProSeal LMA and I-gel LMA, respectively.
  Interventions: Device: endotracheal intubation and laringeal mask airway insertion
- difficult airway manikin with personal protective equipment: The participants will carry out intubation procedure using macintosh direct laryngoscope, GlideScope video laryngoscope, C-Mac video laryngoscope and Frova intubation catheter and laryngeal mask insertion using ProSeal LMA and I-gel LMA, respectively.
  Interventions: Device: endotracheal intubation and laringeal mask airway insertion

INTERVENTIONS:
Device: endotracheal intubation and laringeal mask airway insertion — endotracheal intubation and laringeal mask airway insertion on the airway manikin with different devices

SUMMARY:
Covid-19 disease has caused a worldwide pandemic. However, it was necessary to reduce the transmission of the disease as much as possible. The highest risk of transmission is airway management. Medical personnel responsible for airway management are at the greatest risk. One of the most important ways to protect anesthetists from contamination is to use PPE. But, it should be considered that there is some disadvantage about using PPE. The investigators aimed to evaluate the effects of the use of personal protective equipment and standard uniform during airway management.

DETAILED DESCRIPTION:
Objective: The investigators aimed to compare the effects of the use of personal protective equipment and standard uniform during airway management using direct laryngoscope, GlideScope video laryngoscope, C-Mac video laryngoscope, I-gel laryngeal mask airway , ProSeal laryngeal mask airway and Frova intubation catheter on the manikin that created both difficult airway and normal airway conditions in the Department of Anesthesiology and Reanimation at the Derince Training and Research Hospital, University of Health Sciences.

Materials and Methods: The study will carry out with 24 participants in Health Sciences University Kocaeli Derince Health Education and Research Center. In the study, a simulation manikin will use to evaluate the effect of personal protective equipment use on airway management. Anesthesia technicians, anesthesia residents and specialists will include as participants. As demographic data, the clinical positions of the participants, their experiences with each airway method and the use of personal protective equipment, age, gender, height and weight information will be recorded. Each procedure will be explained to the participants by an anesthesiology specialist and a resident. Then the participants perform their procedure first with standard uniform and then by wearing personal protective equipment. Endotracheal intubation with direct laryngoscope, GlideScope video laryngoscope, C-Mac video laryngoscope and Frova intubation catheter followed by I-gel and ProSeal laryngeal mask airway will be used, respectively. Each procedure will be carried out by creating normal and difficult airway conditions, respectively. Time, number of attempts and presence of optimization maneuver will be recorded for each procedure. Modified CLS (Cormack Lehane Score) and POGO (Percentage Of Glottic Opening) scores will be also recorded during intubation procedures. Each participant will be asked to give a score between 1 and 100 using the Visual Analogue Scale (VAS) in order to evaluate the difficulty of intervention after each procedure subjectively and it will be recorded. Finally, the other subjective effects of personal protective equipment using on participants (such as sweating, feeling of warmth) will be asked.

ELIGIBILITY:
Inclusion Criteria:

* Being an anesthesiology resident, specialist or nurse

Exclusion Criteria:

* Anxiety Disorder
* Severe heart or lung disease
* Claustrophobia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiology residents, anesthesiology specialists or anesthesia nurses will be participants in this study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of times | 2 minutes
  For intubations from holding the laryngoscope to ventilation, for laryngeal mask airway insertion from holding the laryngeal mask airway to ventilation For intubation time from holding the laryngoscope to observing glottic opening for standard uniform.
Evaluation of times | 4 minutes
  For intubations from holding the laryngoscope to ventilation, for laryngeal mask airway insertion from holding the laryngeal mask airway to ventilation For intubation time from holding the laryngoscope to observing the glottic opening for personal protective equipment.
Evaluation of number of attempts | 2 minutes
  For both intubation and laryngeal mask airway insertion, number of attempts until ventilation
Evaluation of presence of optimisation maneuver | 30 seconds
  Whether there is optimisation maneuver for each attempt whether there is maneuver for each attempt
Evaluation of Modified Cormack/Lehane classification | 30 seconds
  The classification includes 5 grades; grade 1, 2a, 2b, 3 and 4. Grade 1 defines the best image of glottis.
Evaluation of Percentage of Glottic Opening Scores | 30 seconds
  Percentage of Glottic Opening describes the percentage of the glottic opening as percentages (0-100). Number 100 describes that the participants see all glottic openings. Number 0 describes that nothing is seen.

SECONDARY OUTCOMES:
Visual Analog Scale of using personal protective equipment | 15 minutes
  The visual analog scale is a scale that converts a subjective property to digital data. It has values between 0-100. Generally it is used for describing pain level. But it is used for describing the difficulty of attempts in this study. Number 0 explains that the attempt is very easy and number 100 is very difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yilmaz, 2, Study Director — University of Healt Sciences, Kocaeli Derince Education and Research Hospital
Locations (1):
- Aydan Okuyucu, Kocaeli, Kocaeli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No